CLINICAL TRIAL: NCT05521659
Title: A Systematic Oral Care Protocol in Non-Mechanically Ventilated Stroke Patients
Brief Title: Oral Care in Non-Mechanically Ventilated Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Bakirkoy Prof. Dr. Mazhar Osman Hospital for Psychiatry, Neurology and Neurosurgery (Unknown)
Responsible Party: Principal Investigator, Zeliha Tülek, Assoc.Prof, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Oral Care in Stroke
Record Dates: First submitted 2022-01-11; First posted 2022-08-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Stroke, Ischemic
Keywords: oral care; stroke; oral mucosa; colonization; bacteria
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standardized oral care protocol (Experimental): Intervention: Patients in experimental group were given oral care 3 times a day at certain hours (06-14-22) with oral care set including chlorhexidine gluconate.
  Interventions: Other: Standardized oral care protocol
- Control Group (No Intervention): Routine oral care (usual oral care with the same appliances and solution but applied twice a day without following a protocol)

INTERVENTIONS:
Other: Standardized oral care protocol — Standardized oral care protocol (3 times a day at certain hours (06-14-22) with oral care set including chlorhexidine gluconate)
  Arms: Standardized oral care protocol

SUMMARY:
This study was conducted to examine the effect of a systematic oral care protocol on bacterial colonization of the oral mucosa in non-mechanically ventilated stroke patients. This experimental study was conducted in Bakirkoy Prof. Dr. Mazhar Osman Research and Training Hospital for Psychiatry, Neurology and Neurosurgery between January -June 2020. The research was carried out with 42 stroke patients who were hospitalized in the intensive care unit but not underwent mechanical ventilation. A standardized oral care protocol was developed and applied to the patients in the experimental group three times a day. The control group underwent non-standardized oral care, which is available in the routine practice of the clinic. Two groups were compared at baseline and at the 5th day of hospital stay in terms of bacterial colonization, oral cavity and complications.

DETAILED DESCRIPTION:
This experimental study was conducted in Bakirkoy Prof. Dr. Mazhar Osman Research and Training Hospital for Psychiatry, Neurology and Neurosurgery between January -June 2020. The research was carried out with 42 stroke patients who were hospitalized in the intensive care unit but not underwent mechanical ventilation. A standardized oral care protocol was developed and applied to the patients in the experimental group three times (at 06:00, 14:00, 22:00) a day (with use of an oral hygiene kit including chlorhexidin gluconate). The control group underwent usual care (oral care with use of the same kit but applied twice a day without following a protocol). Two groups were compared at baseline and at the 5th day of hospital stay in terms of bacterial colonization, oral cavity (by use of Oral Assessment Guide) and complications.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of stroke,
* Being not connected to a mechanical ventilator (patients who were on spontaneous breathing or receiving oxygen support with a mask or nasal cannula),
* Having at least 3 teeth, and
* Cannot meet the need for oral care.

Exclusion Criteria:

* Patients who were intubated or tracheostomized were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
the number of bacteria variable | 5 days.
  The number of bacteria in the oral mucosa of stroke patients who are given oral care according to the standardized oral care protocol after the intervention will be less than the pre-intervention and control groups.

SECONDARY OUTCOMES:
the type of bacteria variable | Evaluation will be done at the beginning of the study and at the end of the 5th day.
  The type of bacteria in the oral mucosa of stroke patients who are given oral care according to the standardized oral care protocol after the intervention will be less than the pre-intervention and control groups.
oral evaluation scale variable | Evaluation will be done at the beginning of the study and at the end of the 5th day.
  The mean Oral Evaluation Scale score of stroke patients who are given oral care according to the standard oral care protocol after the intervention will be lower than the pre-intervention and control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Zeliha Tülek, RN, PhD, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- İstanbul Bakırköy Prof. Dr. Mazhar Osman Ruh Sağlığı ve Sinir Hastalıkları Eğitim ve Araştırma Hastanesi /, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chipps EM, Carr M, Kearney R, MacDermott J, Von Visger T, Calvitti K, Vermillion B, Weber ML, Newton C, St Clair J, Harper D, Yamokoski T, Belcher M, Ali N, Hoet AE, Van Balen J, Holloman C, Landers T. Outcomes of an Oral Care Protocol in Postmechanically Ventilated Patients. Worldviews Evid Based Nurs. 2016 Apr;13(2):102-11. doi: 10.1111/wvn.12124. Epub 2016 Jan 14. PMID 26765505
- [Background] Emery KP, Guido-Sanz F. Oral care practices in non-mechanically ventilated intensive care unit patients: An integrative review. J Clin Nurs. 2019 Jul;28(13-14):2462-2471. doi: 10.1111/jocn.14829. Epub 2019 Mar 13. PMID 30793402